CLINICAL TRIAL: NCT00121602
Title: Randomized, Double-Blind, Equivalence Study of the Efficacy of Darbepoetin Alfa Manufactured by Serum Free Bioreactor Technology and Darbepoetin Alfa Manufactured by Roller-Bottle Technology for the Treatment of Anemia in Patients With Chronic Kidney Disease Receiving Hemodialysis
Brief Title: Efficacy Study: Darbepoetin Alfa for the Treatment of Anemia in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20040104
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Anemia; Kidney Disease
Keywords: Hemodialysis; Darbepoetin Alfa; Clinical Trials; Nephrology; Amgen; Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Anemia; Kidney Diseases; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Roller bottle (Active Comparator)
  Interventions: Drug: Darbepoetin Alfa
- Serum free (Experimental)
  Interventions: Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa — Initial dose, frequency and route of administration of study drug will be the same as that administered for darbepoetin alfa prior to enrollment. Frequency either once a week or once every two weeks, frequency may not change for duration of study. Route of administration either subcutaneous or intravenous, route of administration may not change for duration of study. Study drug provided in pre-filled syringes at the following unit doses: 10, 15, 20, 30, 40, 50, 60, 80, 100 or 150 ug.

SUMMARY:
The purpose of this study is to evaluate whether the efficacy of darbepoetin alfa SF is equivalent to that of darbepoetin alfa RB for the treatment of anemia in patients with chronic kidney disease (CKD) receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of CKD and receiving hemodialysis for greater than or equal to 3 months before enrollment - No prior exposure to EPREX® or NeoRecorman® - Baseline hemoglobin (Hb) between 10 and 13 g/dL - On stable weekly or once every other week intravenous (IV) or subcutaneous (SC) darbepoetin therapy for at least 6 weeks prior to screening (stable is defined as less than 25% change in weekly dose and no change in frequency) - Adequate iron stores (serum ferritin equal to or greater than 100 mg/L) - Before any study-specific procedure, the appropriate written informed consent must be obtained Exclusion Criteria: - Scheduled to receive a kidney transplant - Uncontrolled hypertension, defined as a pre-dialysis systolic blood pressure (BP) greater than 180 and/or diastolic BP of greater than 110 - Acute myocardial ischemia; hospitalization for congestive heart failure, myocardial infarction, deep vein thrombosis, cerebrovascular event (stroke or transient ischemic attack) within 12 weeks before enrollment - Parathyroid hormone (PTH) level greater than 1500 pg/mL - Major surgery within 12 weeks before enrollment (excluding vascular access surgery) - Currently receiving antibiotic therapy for systemic infection - Known positive HIV antibody or positive hepatitis B surface antigen - Clinical evidence of current malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia - Red blood cell (RBC) transfusions within 8 weeks before enrollment - Androgen therapy within 8 weeks before enrollment - Systemic hematologic disease (e.g., sickle cell anemia, myelodysplastic syndromes, hematologic malignancy; myeloma; hemolytic anemia) - Any disorder that may impact (in the judgment of the investigator) the ability to give informed consent for participation in this study - Pregnant or breast-feeding women. All subjects must practice adequate contraception (in the judgment of the investigator) throughout this trial. - Treatment with an investigational agent or device within 30 days before enrollment or scheduled to receive an investigational agent other than those specified by this protocol during the course of this study - Subject has known sensitivity to any of the products to be administered during dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2005-03; Primary Completion 2005-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change in Hb level between the screening/baseline period and the evaluation period | 30 weeks
The ratio of weekly dosing requirements between baseline and the evaluation period | 28 weeks

SECONDARY OUTCOMES:
Change from baseline Hb over time | 29 weeks
Proportion of subjects maintaining mean Hb within target range during evaluation period | 7 weeks
Average darbepoetin alfa dose over evaluation period | 7 weeks
Change from baseline dose over time | 29 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20040104.pdf